CLINICAL TRIAL: NCT04285086
Title: A Phase 3, Open-Label, Multicenter, Randomized, Active-controlled Study to Assess PK and Compare the Efficacy, Safety, and Tolerability of P1101 vs Anagrelide as 2nd Line Therapy for Essential Thrombocythemia (SURPASS ET): The Core Study and Its Extension Study.
Brief Title: Ropeginterferon Alfa-2b (P1101) vs. Anagrelide in Essential Thrombocythemia Patients With Hydroxyurea Resistance or Intolerance
Acronym: SURPASS ET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1101 ET
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Essential Thrombocythemia
Keywords: Essential Thrombocythemia; Ropeginterferon; P1101; PharmaEssentia; MPN; Myeloproliferative neoplasms; ET; JAK2; CALR; MPL; IFN
MeSH Terms: conditions — Thrombocythemia, Essential; Myeloproliferative Disorders | interventions — anagrelide

STUDY DESIGN:
Intervention Model Description: Experimental Drug (Biological): Ropeginterferon alfa-2b (P1101), Q2W, SC injection Control Drug: Anagrelide, capsules, daily, p.o.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropeginterferon alfa-2b (P1101) (Experimental): Pre-filled Syringe, Q2W, SC injection
  Interventions: Biological: Ropeginterferon alfa-2b
- Anagrelide (Active Comparator): Capsules, Daily, p.o.
  Interventions: Drug: Anagrelide

INTERVENTIONS:
Biological: Ropeginterferon alfa-2b — Ropeginterferon alfa-2b (P1101) dosage: from 250 mcg to 500 mcg
  Other Names: P1101
  Arms: Ropeginterferon alfa-2b (P1101)
Drug: Anagrelide — Anagrelide dosage: 0.5 mg per capsule, according to label and physician's judgement
  Arms: Anagrelide

SUMMARY:
This is a Phase 3 open-label, multicenter, randomized, active-controlled study designed to compare the efficacy and safety and tolerability of P1101 compared with ANA after 12 months of treatment as second-line therapy for subjects with ET who have had a suboptimal or failed response to HU.

DETAILED DESCRIPTION:
PharmaEssentia Corporation is developing a pegylated (PEG) IFN-α product, P1101, for the treatment of ET.

Available clinical data and experience with P1101 in PV shows that the compound, with proper dose modifications, is effective in controlling disease in a significant proportion of subjects with ET. Further, its increased serum half-life presents distinct advantages for ET treatment over that of standard IFN-α and other available PEG IFN-α therapy. This pivotal Phase 3 study will establish the efficacy and safety of P1101 in ET subjects.

In core study phase, the enrolled subjects will be randomized into two arms, the test arm is P1101, the control arm is ANA. The overall duration for each eligible patient is 14 months, including screening (1 month), treatment (12 months) and follow-up (1 month) period. Efficacy evaluations, safety assessments, and PK and immunogenicity evaluations of P1101 will be performed.

Evaluation of efficacy will include clinical laboratory assessments, allelic burden measurements of CALR, JAK-2, and MPL, spleen size measurements, bone marrow sampling, EQ-5D-3L, and MPN-SAF TSS completion.

Evaluation of safety will include assessing vital signs, clinical safety laboratory tests, physical examinations, ECG evaluation, heart ECHO, lung X-ray, ECOG performance status, ocular examination, and AEs.

Subjects who completed the end of treatment (EoT) and safety follow-up (EoS) visits of the SURPASS ET study and may benefit from P1101 therapy have the opportunity to receive P1101 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years old
2. Subjects diagnosed with high-risk ET (either older than 60 years and JAK2V617-positive at screening, or having disease-related thrombosis or hemorrhage in the past), diagnosed according to the World Health Organization (WHO) 2016 criteria
3. Subjects have received prior HU for ET, while the washout between the last dose of HU and randomization should not be shorter than 7 days
4. Interferon treatment-naïve, or anti-P1101 binding antibody negative at screening and the washout between last dose of interferon and randomization should not be shorter than 14 days.
5. Documented resistance/intolerance to prior HU for ET, referencing modified ELN criteria (Barosi, et al, 2007), whereby at least one of the following criteria is met:

   Platelet count >600 x 10^9/L at ≥2 g/day (or ≥2.5 g/day if subject body weight >80 kg) or maximally tolerated dose if <2 g/day after at least 3 months of HU, or Platelet count >400 x 10^9/L and WBC count <2.5 x 10^9/L at any dose and any duration of HU, or Platelet count >400 x 10^9/L and hemoglobin (HGB) <10 g/dL at any dose and any duration of HU, or Presence of HU-related toxicities at any dose and any duration of therapy (e.g., leg ulcers, mucocutaneous manifestations, pneumonitis, or HU-related fever), or Platelet count >450 x 10^9/L at any dose and any duration of HU. The actual dose and duration of HU must be recorded on the eCRF. Moreover, if patient received one dose of HU, the reason why subject was judged to be HU resistance/intolerance must be recorded on the eCRF.
6. Platelets >450 x 10^9/L at screening
7. WBC >10 x 10^9/L at screening
8. HGB ≥11 g/dL at screening for males and 10 g/dL at screening for females
9. Neutrophil count ≥1.0 x 10^9/L at screening
10. Adequate hepatic function defined as bilirubin ≤1.5 x upper limit normal (ULN), prothrombin time (PT) (international normalized ratio, INR) ≤1.5 x ULN, albumin >3.5 g/dL, alanine aminotransferase ≤2.0 x ULN, aspartate aminotransferase ≤2.0 x ULN at screening
11. Creatinine clearance ≥40 mL/min (by Cockcroft-Gault equation)
12. Males and females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use an acceptable form of birth control until 28 days following the last dose of the study drug, and females must agree to not breastfeed during the study
13. Written informed consent obtained from the subject and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

1. Any subject requiring a legally authorized representative
2. Any contraindications or hypersensitivity to IFN-α or ANA and their excipients
3. Known risk factors for QT-prolongation (e.g., congenital long QT, known history of acquired QT-prolongations). Medications that can prolong QTc and induce hypokalemia will not be allowed in the study.
4. Co-morbidity with severe or serious condition that, in the Investigator's opinion, would jeopardize the safety of the subject or their compliance with the protocol, including significant cardiac disease (including New York Heart Association Class III-IV congestive heart failure and clinically significant arrhythmias) and pulmonary hypertension
5. History of major organ transplantation
6. Pregnant or lactating females
7. Subjects with any other significant medical conditions that, in the opinion of the Investigator, would compromise the results of the study or may impair compliance with the requirements of the protocol, including but not limited to:

   1. Documented autoimmune disease at screening or in the history (e.g., thyroid dysfunction, hepatitis, idiopathic thrombocytopenic purpura, scleroderma, psoriasis, or any arthritis of autoimmune origin)
   2. Clinically relevant pulmonary infiltrates, pneumonia, and pneumonitis at screening that, in the Investigator's opinion, would jeopardize the safety of the subject or their compliance with the protocol
   3. Infections with systemic manifestations (e.g., bacterial, fungal, or human immunodeficiency virus [HIV], except hepatitis B [HBV] and/or hepatitis C [HCV], at screening)
   4. Evidence of severe retinopathy (e.g., cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension)
   5. History or presence of clinically relevant depression
   6. Previous suicide attempts or at any risk of suicide at screening, in the judgement of the Investigator
   7. History or presence of clinically significant neurologic diseases
   8. History of any malignancy within 5 years (except Stage 0 chronic lymphocytic leukemia, basal cell, squamous cell, and superficial melanoma)
   9. History of alcohol or drug abuse within the last year
   10. History or evidence of any other MPN
   11. History of splenectomy
8. Use of any investigational drug <4 weeks prior to the first dose of study drug or not recovered from effects of prior administration of any investigational agent
9. Subjects with documented ANA resistance or intolerance (see Appendix 8 for definition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood count remission | month 9 and month 12
  platelets ≤400 x 10^9/L AND white blood cells (WBC) <9.5 x 10^9/L
Improvement or non-progression in disease-related signs | month 9 and month 12
  splenomegaly
Large symptoms improvement or maintain non-progression | month 9 and month 12
  based on the Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS)
Absence of hemorrhagic or thrombotic events | month 9 and month 12
  absence of hemorrhagic or thrombotic events

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Sato, MD/PhD, Study Director — PharmaEssentia Japan K.K.; Craig Zimmerman, PhD, Study Director — PharmaEssentia USA Corp.
Locations (65):
- United States (3):
  - Washington University School of Medicine - Division of Oncology, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Canada (3):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (15):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality
  - NanFang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technolog, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital affiliated to Shanghai Jiao Tong University school of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
- Queen Mary Hospital, Hong Kong, Hong Kong
- Japan (13):
  - Ehime University Hospital, Tōon, Ehime
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - University of Miyazaki Hospital, Miyazaki, Miyazaki
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Shizuoka Hospital, Izunokuni, Shizuoka
  - Juntendo University Hospital, Bunkyo City, Tokyo
  - Nippon Medical School Hospital, Bunkyo City, Tokyo
  - NTT Medical Center Tokyo, Shinagawa City, Tokyo
  - Tokyo Medical University Hospital, Shinjuku, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (7):
  - Daegu Catholic University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - SoonChunHyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (21):
  - Chia-Yi Christian Hospital, Chiayi City, Chiayi County
  - Chiayi Chang Gung Memorial Hospital, Chiayi City, Chiayi County
  - Kaohsiung Veterans General Hospital, Kaohsiung City, Kaohsiung City
  - E-Da Cancer Hospital, Kaohsiung City, Kaohsiung City
  - E-Da Hospital, Kaohsiung City, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City, New Taipei City
  - Tainan Municipal An-Nan Hospital, Tainan, Tainan City
  - Chi Mei Medical Center, Tainan, Tainan City
  - Chi-Mei Hospital - Liouying Branch, Tainan, Tainan City
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taipei City
  - Taipei Municipal Wan Fang Hospital, Taipei, Taipei City
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mesa R, Gill H, Zhang L, Jin J, Kirito K, Komatsu N, Qin A, Xiao Z, Tashi T, Shimoda K, Ohishi K, Chen S, Zuo X, Shirane S, Hu Y, Zhang S, Wang Y, Takenaka K, Ichii M, Xu N, Shih LY, Lim KH, Lee SE, Bae SH, Teo WZY, Maze D, Oh ST, Bose P, Sato T, Zagrijtschuk O, Lin S, Shih WJ, Mascarenhas J, Masarova L; SURPASS-ET Study Group. Ropeginterferon alfa-2b in hydroxyurea-intolerant or hydroxyurea-refractory essential thrombocythaemia (SURPASS ET): a multicentre, open-label, randomised, active-controlled, phase 3 study. Lancet Haematol. 2025 Nov;12(11):e862-e875. doi: 10.1016/S2352-3026(25)00264-9. PMID 41193116
- [Derived] Verstovsek S, Komatsu N, Gill H, Jin J, Lee SE, Hou HA, Sato T, Qin A, Urbanski R, Shih W, Zagrijtschuk O, Zimmerman C, Mesa RA. SURPASS-ET: phase III study of ropeginterferon alfa-2b versus anagrelide as second-line therapy in essential thrombocythemia. Future Oncol. 2022 Sep;18(27):2999-3009. doi: 10.2217/fon-2022-0596. Epub 2022 Aug 4. PMID 35924546